CLINICAL TRIAL: NCT04663334
Title: Change in Coronary Microcirculation and Fractional Flow Reserve After Transcatheter Aortic Valve Implantation in Patients With Concomitant Coronary Artery Disease and Severe Aortic Stenosis.
Brief Title: Change in Coronary Microcirculation and FFR After TAVI in Patients With Cardiovascular Comorbidities
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: AP001
Record Dates: First submitted 2020-12-04; First posted 2020-12-11 (Actual); Last update posted 2023-12-15 (Actual); Status verified 2023-12

CONDITIONS: Severe Symptomatic Aortic Stenosis
Keywords: Coronary Flow Reserve; Index of Microvascular Resistance; Fractional Flow Reserve; Transcatheter Aortic Valve Implantation; Coronary Artery Disease; Severe Aortic Stenosis
MeSH Terms: conditions — Coronary Artery Disease; Aortic Valve Stenosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: inverse myocardial remodeling — a myocardial reverse remodeling is described, generating a decrease in hypertrophy, interstitial oedema, and inflammation. Its effect on coronary microcirculatory reserve is not known. Some studies have shown improvement in coronary reserve immediately after TAVI and this effect seemed to last long after treatment

SUMMARY:
Change in coronary microcirculation and Fractional Flow Reserve after Transcatheter Aortic Valve Implantation in patients with concomitant coronary artery disease and severe aortic stenosis.

Severe aortic stenosis is the most common indication of valvular replacement in developed countries. Stable coronary artery disease (CAD) is frequently associated with severe aortic stenosis in patients treated by Transcatheter Aortic Valvular Implantation (TAVI). Its prognostic impact is not clearly established, and available studies uncommonly used functional assessment of severity from a coronary stenosis to stratify the risk in this situation.

Fractional Flow Reserve (FFR) is recommended to guide revascularization by percutaneous coronary intervention (PCI) in clinical practice. Its use is not validated in patients with severe aortic stenosis. Left ventricular hypertrophy induced by aortic obstruction leading to microvascular disorders, and can alter coronary reserve, possibly biasing FFR values. After aortic valvular replacement, a myocardial reverse remodeling is described, generating a decrease in hypertrophy, interstitial oedema, and inflammation. Its effect on coronary microcirculatory reserve is not known. Some studies have shown improvement in coronary reserve immediately after TAVI and this effect seemed to last long after treatment.

The aim of the study is to assess the effects of inverse myocardial remodeling on coronary microcirculatory function and its association with FFR values before and after TAVI.

DETAILED DESCRIPTION:
This monocentric and prospective observational study aims to include patients with stable coronary artery disease and undergoing TAVI for severe aortic stenosis via transfemoral access, from November 2020 at Nantes University Hospital, France.

All patients have severe symptomatic aortic stenosis, secondary to degenerative disease confirmed by transthoracic echocardiography (mean gradient >40 mmHg and/or valve area <1 cm2) and significant epicardial coronary stenosis (> or = 50%) assessed by coronarography performed in systematic preoperative work-up. These patients are deemed for TAVI and a first-line medical treatment for CAD, after heart team decision.

The collegially chosen strategy to manage CAD in this population consists in assessing hemodynamic parameters from a coronary stenosis during the TAVI procedure, using functionals tests for ischemia (FFR, IMR, CFR) from a concomitant coronarography. Patients will be routinely admitted in hospital 6 months after TAVI, for clinical and echocardiographic reassessment, and coronarography control. Functional tests will be repeated and according to results, continuation of medical therapy or PCI is proposed, at operator's discretion.

All procedures are performed within the same site by 1 medical team including 4 interventional cardiologists.

Before the TAVI procedure, a computerized multi-sliced tomography is systematically performed to validate the percutaneous approach by femoral access and to choose which prothesis model will be used.

In most cases, TAVI procedure are performed under local anesthesia and mild sedation, under anesthetist supervision.

The common femoral artery is punctured by percutaneous approach, above the femoral bifurcation and a 16-French sheath is inserted.

Three available models of aortic bioprothesis are implanted in our center, the Sapien 3 (EDWARDS Lifescience) the Corevalve Evolute R (Metdtronik) and the Accurate Neo 2 (Boston Scientific) Two Perclose ProGlide devices (Abbott Vascular) are used to perform the perpendicular preclosing. After the deployment of the prosthesis, the TAVI sheath is removed and the nodes from the two previously placed ProGlide devices are tightened. Final femoral angiographic control is not systematic.

Concomitant coronarography is performed by radial artery access site, using a 6-French sheath.

Hemodynamics measures are recorded by PressureWire X Guidewire (Abott Vascular) wireless devices to a computer and processed by the CoroFlow Coroventis software (Abbott Vascular) to carry out multimodal physiological evaluation. FFR, CFR, and IMR measures will be repeated before and immediately after valve implantation. These parameters will be reassessed 6 months after TAVI.

ELIGIBILITY:
Inclusion Criteria:

* Adults older than 18 years. For female of childbearing age, active contraceptive method is recommended.
* patients with severe symptomatic aortic stenosis secondary to degenerative disease confirmed by transthoracic echocardiography (mean gradient >40 mmHg and/or valve area <1 cm2) and with significant coronary artery disease (epicardial coronary stenosis angiography > or = to 50%)

Exclusion Criteria:

* Severe CAD with tritroncular lesions or severe stenosis (>90 %) of left main artery or proximal left anterior descending artery

  * Lack of viability in myocardial territory of interest
  * History of bypass coronary surgery or heart transplantation
  * Severe left ventricular systolic dysfunction, characterized by an ejection fraction < 35 %
  * Severe renal impairment (Creatinine clearance <30 ml/min/1.73 m2)
  * Absolute contraindication to intravenous adenosin
  * Pregnant or nursing women Patients under guardianship, curatorship, or protection of justice

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients have severe symptomatic aortic stenosis, secondary to degenerative disease confirmed by transthoracic echocardiography (mean gradient >40 mmHg and/or valve area <1 cm2) and significant epicardial coronary stenosis (> or = 50%) assessed by coronarography performed in systematic preoperative work-up. These patients are deemed for TAVI and a first-line medical treatment for CAD, after heart team decision.
Sampling Method: Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2020-12-08 (Actual); Primary Completion 2023-05-08 (Actual); Study Completion 2023-05-08 (Actual)

PRIMARY OUTCOMES:
Study the change in FFR values before and 6 months after TAVI | 6 months
  FFR values are presented as median and interquartile range. FFR values comparisons pre-TAVI, post-TAVI, and 6 month after procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Thierry Manigold, Study Director — Nantes University Hospital
Locations (1):
- CHU Nantes, Nantes, France

REFERENCES:
- [Derived] Battistolo Q, Le Ruz R, Piriou PG, Guerin P, Letocart V, Plessis J, Poinas A, Senage T, Manigold T. Changes in microcirculation following transcatheter aortic valve implantation in patients with stable coronary artery disease. Arch Cardiovasc Dis. 2025 Apr;118(4):222-230. doi: 10.1016/j.acvd.2024.12.006. Epub 2024 Dec 21. PMID 39827054